CLINICAL TRIAL: NCT03146806
Title: Safety of Intranasal Ketamine for Reducing Uncontrolled Cancer Related Pain
Brief Title: Intranasal (NAS) Ketamine for Cancer Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Vinita Singh, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00086610
Record Dates: First submitted 2017-05-03; First posted 2017-05-10 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Cancer; Pain
Keywords: Cancer pain; Anesthesiology; Opiates; Intranasal ketamine
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intranasal ketamine treatment (Experimental): Study participants who are receiving intranasal ketamine treatments.
  Interventions: Drug: Intranasal ketamine

INTERVENTIONS:
Drug: Intranasal ketamine — 10mg of intranasal ketamine will be given to make sure that the study patients are able to tolerate a small dose of NAS ketamine.
  On the second visit, 10 mg of IV ketamine will be given to help establish bioavailability of NAS ketamine, with patients serving as their own controls.
  On the third and fourth visit, higher doses of ketamine, 30 mg and 50 mg respectively, will be given.
  All doses of ketamine will be administered by an anesthesia research nurse.
  Other Names: NAS ketamine; Ketamine hydrochloride (HCl) intranasal

SUMMARY:
The main purpose of this study is to determine the safety, feasibility, and utility of intranasal (NAS) ketamine in persistent uncontrolled cancer related pain. In this prospective clinical trial the researchers will investigate the use of NAS ketamine in patients with pain related to cancer or cancer treatment. The researchers plan to enroll at least 25 patients meeting inclusion/exclusion criteria, to achieve a minimum of 10 patients who complete the study. Participants will be recruited from the supportive oncology clinic, oncology clinics, the pain clinic and Acute Pain Service at Emory. Participants will be asked to return to the Phase I unit of the Winship Cancer Building C for a total of 5 study visits, each two to five days apart. During these visits participants will complete questionnaires, have blood samples drawn and will have study medication administered to them in escalating doses. For safety monitoring participants will be contacted by telephone 14 days after the last dose of medication administered.

DETAILED DESCRIPTION:
There are about 11.9 million Americans affected with cancer. 53% of patients with cancer experience pain at all stages of cancer. These patients often require high doses of opioids with uncontrolled pain that makes them too sedated to effectively participate in day-to-day activities and have a good quality of life. Depression often co-exists with cancer pain due to the nature of the disease. The researchers are searching for improved therapies for chronic cancer pain and ketamine with its novel mechanism of action may be a promising solution.

Ketamine is an FDA approved anesthetic with the ability to effect memory loss, pain relief and sedation. Safety and efficacy of ketamine as an anesthetic and analgesic agent is well documented. Low doses of ketamine have minimal adverse impact on circulatory or breathing functions but can reduce pain. Research has shown that ketamine is effective in controlling breakthrough pain and reducing depression in a randomized double blind controlled trial. There is limited data regarding the use of ketamine for pain management in cancer.

One of the challenges with ketamine is the route of administration, most commonly given intravenously (IV) or intramuscularly (IM). It has also been given by mouth and rectally, but absorption is very poor. Intranasal (NAS) administration may be a promising method of delivery and can be ordered by a physician from a compounding pharmacy. From other research the investigators expect absorption to be higher than oral or rectal administration and this method of delivery as needle-free is a patient-friendly route of administration.

The main purpose of this study is to determine the safety, feasibility, and utility of intranasal (NAS) ketamine in persistent uncontrolled cancer related pain. In this prospective clinical trial the researchers will investigate the use of NAS ketamine in patients with pain related to cancer or cancer treatment. The researchers plan to enroll at least 15 patients meeting inclusion/exclusion criteria, to achieve a minimum of 10 patients who complete the study. Participants will be recruited from the oncology clinic, pain clinic and Acute Pain Service at Emory. Participants will be asked to return to the Phase I unit of the Winship Cancer Building C for a total of 5 study visits, each two to five days apart. During these visits participants will complete questionnaires, have blood samples drawn and will have study medication administered to them in escalating doses. For safety monitoring participants will be contacted by telephone 14 days after the last dose of medication administered.

Data obtained from this study will help determine if ketamine provides a reduction of pain using the Numeric Pain Rating Scale and a reduction in the use of opioid consumption and other rescue medications. Additionally the researchers will study the bioavailability, pharmacodynamics and pharmacokinetics of ketamine and the safety profile of NAS ketamine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncontrolled pain related to cancer or cancer treatment. Uncontrolled pain will be defined as:

  * Pain which persists for more than 7 days and is rated >/=4 on Numerical Pain Rating Score (NPRS)
  * Use of breakthrough medication more than 4 times in 24 hours or being treated with oral morphine equivalent of 50 mg/d or more
* Patients who are able to follow-up in person during the trial
* Patient on stable analgesic regimen for >7 days without escalation during study period with rescue or immediate release medication every 3 hours or longer
* Patients who are willing and able to maintain a daily pain diary
* Patients who are able to understand written and verbal English
* Patient weight >/= 50 kg

Exclusion Criteria:

* Transportation issues interfering with return study visits
* Patients with high disposition of laryngospasm or apnea
* Presence of severe cardiac disease
* Presence of conditions where significant elevations in blood pressure would be a serious hazard.
* Stage 2 hypertension or greater (systolic blood pressure > 160 and/or diastolic blood pressure >100)
* Baseline tachycardia, heart rate (HR) >100
* History of seizures, elevated intracranial pressure (ICP) or cerebrospinal fluid (CSF) obstructive states (e.g. severe head injury, central congenital or mass lesions)
* Conditions that may increase intraocular pressure (e.g. glaucoma, acute globe injury)
* History of uncontrolled depression or other psychiatric comorbidity with psychosis
* History of liver disease
* History of interstitial cystitis
* History of nasal or sinus anomalies or dysfunction e.g. allergic or infectious rhinitis.
* Patients with lesions to the nasal mucosa
* Pregnant women, nursing mothers and women of childbearing potential not using contraception known to be highly effective. Highly effective contraception methods include combination of any two of the following:

  * Use of oral, injected or implanted hormonal methods of contraception or;
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS);
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
  * Total abstinence or;
  * Male/female sterilization.
* Illicit substance abuse within the past 6 months
* Documented history of medication abuse/misuse (e.g. Unsanctioned dose escalation, broken opioid agreement etc.)
* Clinical requirement for medications that are concurrent inducers or inhibitors of CYP3A4. CYP3A4 substrates are allowed.
* Porphyria (possibility of triggering a porphyric reaction)
* Severe active anemia ( a hemoglobin< 8 documented by labs drawn within 3 months of first study treatment)
* History of difficult intravenous access
* Intractable vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinita Singh, MD, Principal Investigator — Emory University
Locations (1):
- Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shteamer JW, Harvey RD, Spektor B, Curseen K, Egan K, Chen Z, Gillespie TW, Sniecinski RM, Singh V. Safety of Intranasal Ketamine for Reducing Uncontrolled Cancer-Related Pain: Protocol of a Phase I/II Clinical Trial. JMIR Res Protoc. 2019 Apr 30;8(4):e12125. doi: 10.2196/12125. PMID 31038469

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited from the supportive oncology clinic, oncology clinics, and pain clinics at Emory University in Atlanta, Georgia. Participant enrollment began July 25, 2017 and all follow up was complete by April 22, 2020.
Groups:
- Ketamine Treatment: On the first study visit, 10mg of intranasal ketamine was given to make sure that the study patients could tolerate a small dose of intranasal ketamine. On the second visit, 10 mg of intravenous (IV) ketamine was given to compare the two routes of ketamine administration, with patients serving as their own controls. On the third and fourth visit, higher doses of intranasal ketamine, 30 mg and 50 mg respectively, were given, if the patients did not have severe adverse events with the smaller dosage. Participants returned for a fifth visit, 24 hours after Visit 4, to provide a blood sample and complete questionnaires.
Period: Overall Study
Arm/Group | Ketamine Treatment
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intranasal Ketamine Treatment: Study participants receiving three different doses of intranasal ketamine and one dose of IV ketamine, at four different study visits, for treatment of cancer pain.
Arm/Group | Intranasal Ketamine Treatment
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49.5 [31 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Cancer Type [Count of Participants; unit: Participants]
  Breast | 4
  Bone | 2
  Lung | 1
  Colon | 1
  Larynx | 1
  Multiple myeloma | 1
Pain Type [Count of Participants; unit: Participants]
  Nociceptive | 5
  Neuropathic | 0
  Mixed nociceptive and neuropathic pain | 5

OUTCOME MEASURES:

1. Primary Outcome: Bioavailability of Ketamine
Description: Blood samples were obtained at the study visits where ketamine was administered to measure the bioavailability (a pharmacokinetic characteristic) of intranasal and intravenous ketamine. Bioavailability is assessed as nanograms per milliliter (ng/mL) of ketamine circulating in blood. Each study participant received each dose of ketamine during separate study visits. Samples were obtained prior to ketamine administration, and at 2, 30, 60 and 240 minutes after medication administration, during study visits 1 through 4. The baseline sample was not collected at the first study visit as assessing prior intake of ketamine was not necessary.
Time Frame: Baseline, Minutes 2, 30, 60, and 240 during Study Visits 1 through 4, up to 4 weeks
Population: The baseline measurement was not collected during the visit where 10 mg of intranasal ketamine was administered. This analysis includes participants with viable samples. Some samples were not able to be reliably analyzed for this outcome.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- 10 mg Intranasal Ketamine: Study participants receiving 10 mg of intranasal ketamine.
- 10 mg Intravenous (IV) Ketamine: Study participants receiving 10 mg of ketamine intravenously.
- 30 mg Intranasal Ketamine: Study participants receiving 30 mg of intranasal ketamine.
- 50 mg Intranasal Ketamine: Study participants receiving 50 mg of intranasal ketamine.
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 7 | 9 | 10 | 10
ng/mL
  Baseline: number analyzed (Participants) | 0 | 9 | 10 | 10
  Baseline |  | 0 (0) | 0 (0) | 0 (0)
  2 minutes post-ketamine administration | 13.4 (1.65) | 296.4 (1.71) | 23.7 (2.98) | 33.7 (3.86)
  30 minutes post-ketamine administration | 20.3 (2.01) | 35.0 (1.35) | 48.6 (1.67) | 51.0 (1.75)
  60 minutes post-ketamine administration | 11.7 (1.38) | 16.4 (1.70) | 26.5 (2.1) | 55.8 (2.12)
  240 minutes post-ketamine administration | 0 (0) | 0 (0) | 0 (0) | 0 (0)

2. Primary Outcome: Peak Concentration (Cmax) of Ketamine
Description: Blood samples were obtained at the study visits where ketamine was administered to measure the peak concentration (Cmax) of intranasal and intravenous ketamine. Peak concentration is assessed as the maximum ng/mL of ketamine circulating in blood. Each study participant received each dose of ketamine during separate study visits. Samples were obtained at 2, 30, 60 and 240 minutes after medication administration.
Time Frame: Minute 2 through Minute 240 during Study Visits 1 through 4, up to 4 weeks
Population: This analysis includes participants with viable samples. Some samples were not able to be reliably analyzed for this outcome.
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 7 | 9 | 10 | 10
ng/ml | 22.9 (1.97) | 296 (1.71) | 60.8 (1.90) | 77.6 (2.29)

3. Primary Outcome: Area Under the Curve of Ketamine
Description: Blood samples were obtained at the study visits where ketamine was administered to measure the elimination (a pharmacokinetic characteristic) of intranasal and intravenous ketamine. Elimination of the drug disappearing from the body is assessed as the area under the curve (AUC). Each study participant received each dose of ketamine during separate study visits. Samples were obtained at 2, 30, 60 and 240 minutes after medication administration. Each subject did not have quantitative levels at all time points. There were not enough data to construct a curve for each participant and therefore calculate an AUC. Data from all participants were naively pooled to calculate one AUC for the entire population (i.e., across all participants' data).
Time Frame: Minute 2 through Minute 240 during Study Visits 1 through 4, up to 4 Weeks
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: micrograms•hour/Liter (µg•h/L)
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 7 | 9 | 10 | 10
micrograms•hour/Liter (µg•h/L) | 19 (NA) — Data were naively pooled and the AUC for individual participants was not determined, thus a measure of dispersion is not calculable. | 113 (NA) — Data were naively pooled and the AUC for individual participants was not determined, thus a measure of dispersion is not calculable. | 46 (NA) — Data were naively pooled and the AUC for individual participants was not determined, thus a measure of dispersion is not calculable. | 64 (NA) — Data were naively pooled and the AUC for individual participants was not determined, thus a measure of dispersion is not calculable.

4. Primary Outcome: Time to Peak Concentration (Tmax) of Ketamine
Description: Blood samples were obtained at the study visits where ketamine was administered to measure the time to peak concentration (Tmax) of intranasal and intravenous ketamine. Time is measured as minutes after administration when the maximum concentration of ketamine in blood is reached.
Time Frame: Minute 2 through Minute 240 during Study Visits 1 through 4, up to 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 7 | 9 | 10 | 10
minutes | 23 (3.0) | 2 (1) | 14 (3.8) | 16 (4.4)

5. Primary Outcome: Numerical Pain Rating Scale (NPRS) Score
Description: The Numerical Pain Rating Scale (NPRS) was used to evaluate patient reported pain. Pain scores were recorded prior to and at 5,10,15, 30, 45, 60, 120, 180 and 240 minutes after administration of ketamine. The NPRS asks participants rate their current level of pain intensity on a scale from 0 (no pain) to 10 (worst possible pain). In general, improvements of pain severity of 1.5 points or less on NPRS could be seen as clinically irrelevant. Above that value, the cutoff point for "clinical relevance" depends on patients' baseline pain severity, and ranges from 2.4 to 5.3. Higher baseline scores require larger raw changes to represent clinically important differences.
Time Frame: Baseline, Minutes 5, 10, 15, 30, 45, 60, 120, 180, and 240 during Study Visits 1 through 4, up to 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 7.5 [6 to 8] | 6 [5 to 8] | 5.5 [5 to 7] | 6 [6 to 8]
  Minute 5 | 6 [5 to 8] | 1 [0 to 3] | 5 [4 to 6] | 5 [3 to 5]
  Minute 10 | 6 [5 to 8] | 0 [0 to 3] | 3 [3 to 6] | 4 [2 to 5]
  Minute 15 | 5 [4 to 7] | 1.5 [0 to 3] | 3.5 [3 to 6] | 3 [2 to 5]
  Minute 30 | 4.5 [2 to 7] | 2.5 [0 to 5] | 3.5 [2 to 6] | 2 [2 to 5]
  Minute 45 | 5 [3 to 7] | 3 [0 to 5] | 3 [2 to 4] | 2 [2 to 4]
  Minute 60 | 4.5 [3 to 6] | 3.5 [1 to 5] | 2.5 [2 to 3] | 2 [1 to 5]
  Minute 120 | 4.5 [3 to 7] | 3.5 [1 to 4] | 3 [2 to 3] | 2 [1 to 5]
  Minute 180 | 5 [3 to 6] | 4 [1 to 5] | 3 [2 to 3] | 2.5 [1 to 6]
  Minute 240 | 5 [3 to 7] | 3 [1 to 4] | 3 [3 to 4] | 5 [2 to 6]

6. Primary Outcome: Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) Fatigue Score
Description: To evaluate self-reported fatigue, participants completed the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). During visits 1 through 4, side effects were documented by SERSDA prior to administration of medication and 30, 60 and 240 minutes after ketamine administration. Participants indicated the severity of this side effect by selecting 0 (side effect is absent), 1 (weak side effect), 2 (modest side effect), 3 (bothersome side effect), or 4 (side effect is very bothersome).
Time Frame: Baseline, Minutes 30, 60, and 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 2.9 (0.86) | 1.4 (0.84) | 1.6 (0.70) | 1.5 (1.27)
  Minute 30 | 1 (1.15) | 1.6 (1.17) | 1.3 (1.06) | 1.0 (1.25)
  Minute 60 | 0.7 (0.95) | 1.2 (1.23) | 1.2 (1.14) | 1.2 (1.03)
  Minute 240 | 0.8 (0.92) | 1 (0.82) | 0.8 (1.03) | 0.7 (0.67)

7. Primary Outcome: Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) Dizziness Score
Description: To evaluate self-reported dizziness, participants completed the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). During visits 1 through 4, side effects were documented by SERSDA prior to administration of medication and 30, 60 and 240 minutes after ketamine administration. Participants indicated the severity of this side effect by selecting 0 (side effect is absent), 1 (weak side effect), 2 (modest side effect), 3 (bothersome side effect), or 4 (side effect is very bothersome).
Time Frame: Baseline, Minutes 30, 60, and 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 0.6 (0.97) | 0.1 (0.32) | 0 (0) | 0 (0)
  Minute 30 | 0.1 (0.32) | 0.8 (1.14) | 0.3 (0.67) | 0.5 (0.71)
  Minute 60 | 0 (0) | 0.3 (0.95) | 0.1 (0.32) | 0.2 (0.63)
  Minute 240 | 0 (0) | 0 (0) | 0 (0) | 0 (0)

8. Primary Outcome: Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) Nausea Score
Description: To evaluate self-reported nausea, participants completed the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). During visits 1 through 4, side effects were documented by SERSDA prior to administration of medication and 30, 60 and 240 minutes after ketamine administration. Participants indicated the severity of this side effect by selecting 0 (side effect is absent), 1 (weak side effect), 2 (modest side effect), 3 (bothersome side effect), or 4 (side effect is very bothersome).
Time Frame: Baseline, Minutes 30, 60, and 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 0.2 (0.42) | 0.3 (0.67) | 0.1 (0.32) | 0.1 (0.32)
  Minute 30 | 0.3 (0.95) | 0.8 (1.32) | 0.4 (0.97) | 0.3 (0.67)
  Minute 60 | 0.2 (0.63) | 0.6 (1.07) | 0.1 (0.32) | 0.3 (0.67)
  Minute 240 | 0.1 (0.32) | 0 (0) | 0.4 (0.97) | 0.4 (1.26)

9. Primary Outcome: Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) Headache Score
Description: To evaluate self-reported headache, participants completed the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). During visits 1 through 4, side effects were documented by SERSDA prior to administration of medication and 30, 60 and 240 minutes after ketamine administration. Participants indicated the severity of this side effect by selecting 0 (side effect is absent), 1 (weak side effect), 2 (modest side effect), 3 (bothersome side effect), or 4 (side effect is very bothersome).
Time Frame: Baseline, Minutes 30, 60, and 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 0.2 (0.63) | 0 (0) | 0 (0) | 0 (0)
  Minute 30 | 0 (0) | 0.1 (0.32) | 0 (0) | 0 (0)
  Minute 60 | 0 (0) | 0.1 (0.32) | 0 (0) | 0 (0)
  Minute 240 | 0 (0) | 0 (0) | 0 (0) | 0 (0)

10. Primary Outcome: Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) Feeling of Unreality Score
Description: To evaluate self-reported feeling of unreality, participants completed the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). During visits 1 through 4, side effects were documented by SERSDA prior to administration of medication and 30, 60 and 240 minutes after ketamine administration. Participants indicated the severity of this side effect by selecting 0 (side effect is absent), 1 (weak side effect), 2 (modest side effect), 3 (bothersome side effect), or 4 (side effect is very bothersome).
Time Frame: Baseline, Minutes 30, 60, and 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 0.2 (0.63) | 0 (0) | 0 (0) | 0 (0)
  Minute 30 | 0.4 (1.26) | 1.3 (1.42) | 0.2 (0.42) | 0.2 (0.42)
  Minute 60 | 0 (0) | 0.5 (1.27) | 0 (0) | 0.1 (0.32)
  Minute 240 | 0 (0) | 0.2 (0.63) | 0 (0) | 0 (0)

11. Primary Outcome: Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) Change in Hearing Score
Description: To evaluate self-reported change in hearing, participants completed the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). During visits 1 through 4, side effects were documented by SERSDA prior to administration of medication and 30, 60 and 240 minutes after ketamine administration. Participants indicated the severity of this side effect by selecting 0 (side effect is absent), 1 (weak side effect), 2 (modest side effect), 3 (bothersome side effect), or 4 (side effect is very bothersome).
Time Frame: Baseline, Minutes 30, 60, and 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 0 (0) | 0 (0) | 0.1 (0.32) | 0 (0)
  Minute 30 | 0 (0) | 0.1 (0.32) | 0 (0) | 0 (0)
  Minute 60 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Minute 240 | 0 (0) | 0.3 (0.95) | 0 (0) | 0 (0)

12. Primary Outcome: Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) Change in Vision Score
Description: To evaluate self-reported change in vision, participants completed the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). During visits 1 through 4, side effects were documented by SERSDA prior to administration of medication and 30, 60 and 240 minutes after ketamine administration. Participants indicated the severity of this side effect by selecting 0 (side effect is absent), 1 (weak side effect), 2 (modest side effect), 3 (bothersome side effect), or 4 (side effect is very bothersome).
Time Frame: Baseline, Minutes 30, 60, and 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 0.4 (0.70) | 0.1 (0.32) | 0.1 (0.32) | 0 (0)
  Minute 30 | 0.1 (0.32) | 0.5 (0.85) | 0.1 (0.32) | 0.1 (0.21)
  Minute 60 | 0 (0) | 0.1 (0.32) | 0 (0) | 0.1 (0.32)
  Minute 240 | 0 (0) | 0 (0) | 0 (0) | 0 (0)

13. Primary Outcome: Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) Mood Change Score
Description: To evaluate self-reported mood change, participants completed the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). During visits 1 through 4, side effects were documented by SERSDA prior to administration of medication and 30, 60 and 240 minutes after ketamine administration. Participants indicated the severity of this side effect by selecting 0 (side effect is absent), 1 (weak side effect), 2 (modest side effect), 3 (bothersome side effect), or 4 (side effect is very bothersome).
Time Frame: Baseline, Minutes 30, 60, and 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 0.5 (0.85) | 0 (0) | 0 (0) | 0.5 (1.08)
  Minute 30 | 0 (0) | 0.6 (1.26) | 0.1 (0.32) | 0.4 (0.70)
  Minute 60 | 0 (0) | 0.4 (1.26) | 0 (0) | 0.1 (0.32)
  Minute 240 | 0 (0) | 0 (0) | 0 (0) | 0.3 (0.67)

14. Primary Outcome: Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) General Discomfort Score
Description: To evaluate self-reported general discomfort, participants completed the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). During visits 1 through 4, side effects were documented by SERSDA prior to administration of medication and 30, 60 and 240 minutes after ketamine administration. Participants indicated the severity of this side effect by selecting 0 (side effect is absent), 1 (weak side effect), 2 (modest side effect), 3 (bothersome side effect), or 4 (side effect is very bothersome).
Time Frame: Baseline, Minutes 30, 60, and 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 1.6 (1.51) | 1.3 (1.34) | 1.2 (1.32) | 1.1 (1.45)
  Minute 30 | 0.9 (1.37) | 1.1 (1.45) | 0.8 (1.32) | 0.8 (1.14)
  Minute 60 | 0.6 (1.35) | 0.8 (1.32) | 0.8 (1.32) | 0.8 (1.32)
  Minute 240 | 0.5 (1.08) | 0.8 (1.32) | 0.8 (1.32) | 1.2 (1.62)

15. Primary Outcome: Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) Hallucinations Score
Description: To evaluate self-reported hallucinations, participants completed the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). During visits 1 through 4, side effects were documented by SERSDA prior to administration of medication and 30, 60 and 240 minutes after ketamine administration. Participants indicated the severity of this side effect by selecting 0 (side effect is absent), 1 (weak side effect), 2 (modest side effect), 3 (bothersome side effect), or 4 (side effect is very bothersome).
Time Frame: Baseline, Minutes 30, 60, and 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Minute 30 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Minute 60 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Minute 240 | 0 (0) | 0 (0) | 0 (0) | 0 (0)

16. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) Score
Description: Depression was assessed on the Montgomery Asberg Depression Rating Scale (MADRS) during each study visit, before medication administration and 180 minutes after medication administration. The MADRS is designed to be particularly sensitive to treatment effects. The MADRS is a 10-item scale where the survey administrator rates the participant on a variety of aspects related to depression (such as apparent sadness, tension, and pessimistic thoughts) based on a clinical interview. Responses are provided on a scale of 0 to 6 where 0 signifies no difficulties in this area and 6 signifies severe difficulty. Total scores range from 0 to 60 with higher scores indicating greater severity of depression.
Time Frame: Baseline and Minute 180, during Study Visits 1 through 5, up to 6 weeks
Population: The MADRS assessment was only given at the baseline time point during the follow-up visit as no medication was administered during this visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Follow-up Visit: Participants returned for a fifth visit to complete questionnaires. No study medication was administered during this visit.
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine | Follow-up Visit
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
score on a scale
  Baseline | 18.7 (6.57) | 13.4 (6.40) | 12 (5.05) | 11.89 (8.34) | 14.78 (7.31)
  Minute 180: number analyzed (Participants) | 10 | 10 | 10 | 10 | 0
  Minute 180 | 13.5 (4.38) | 13.3 (5.31) | 11.3 (6.15) | 9.67 (8.34) |

17. Primary Outcome: Edmonton Symptom Assessment System (ESAS) Score
Description: The Edmonton Symptom Assessment System (ESAS) assesses nine symptoms that are common in cancer patients: pain, tiredness, drowsiness, nausea, lack of appetite, shortness of breath, depression, anxiety, and well-being. Each symptom is rated on a scale ranging from 0 (absence of symptom) to 10 (worst possible degree of symptom). The ESAS was administered at the baseline time point at each study visit.
Time Frame: Baseline during Study Visits 1 through 5, up to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine | Follow-up Visit
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
units on a scale
  Pain | 6.64 (1.96) | 6.27 (2.10) | 5.80 (1.81) | 5.73 (2.53) | 5.30 (1.89)
  Tiredness | 6.09 (1.92) | 4.73 (2.57) | 4.20 (2.44) | 4.36 (2.54) | 3.60 (2.11)
  Drowsiness | 4.64 (2.98) | 3.64 (2.58) | 2.90 (2.60) | 3.64 (2.50) | 2.00 (2.21)
  Nausea | 1.09 (2.59) | 0.82 (1.60) | 0.40 (0.70) | 0.227 (0.65) | 0 (0)
  Lack of Appetite | 4.55 (2.77) | 3.45 (2.38) | 3.00 (3.02) | 2.20 (2.10) | 2.20 (2.20)
  Shortness of Breath | 1.55 (2.70) | 1.09 (1.97) | 0.40 (1.26) | 0.18 (0.60) | 0.60 (0.97)
  Depression | 3.18 (2.44) | 2.45 (1.86) | 1.50 (1.51) | 0.82 (1.33) | 2.10 (3.41)
  Anxiety | 3.82 (2.82) | 2.82 (1.94) | 1.00 (1.25) | 1.27 (1.68) | 0.60 (0.97)
  Well-being | 4.82 (2.52) | 4.45 (2.88) | 4.20 (2.20) | 4.09 (2.66) | 4.60 (2.27)

18. Primary Outcome: Eastern Cooperative Oncology Group (ECOG) Score
Description: The Eastern Cooperative Oncology Group (ECOG) score evaluates performance status of the participants by rating their ability to perform physical tasks and self care. Responses are 0 (fully active), 1 (restricted in physical strenuous activity but ambulatory), 2 (ambulatory and capable of all self-care but unable to carry out work activities), 3 (capable of only limited self-care), 4 (completely disabled), or 5 (dead). The ECOG score will be obtained at the baseline time point at each study visit where medication is administered.
Time Frame: Baseline during Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale | 2.1 (0.88) | 2.1 (0.88) | 1.8 (0.79) | 1.9 (0.99)

19. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Score
Description: The PROMIS Global Health questionnaire, version 1.1, consists of 10 items assessing general domains of health and functioning. Items are scored on a 5-point scale where 1 = poor and 5 = excellent. Total scores are standardized to a T-score with a mean of 50 and a standard deviation of 10. Scores above 50 indicate better health and functioning, while scores below 50 indicate physical, mental and social health that is below average.
Time Frame: Baseline during Visit 1 and Visit 5, up to 6 weeks
Population: One participant did not complete the PROMIS questionnaire at the Follow-up Visit.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Visit 1 (10 mg Intranasal Ketamine Administered): Study participants receiving 10 mg of intranasal ketamine.
Arm/Group | Visit 1 (10 mg Intranasal Ketamine Administered) | Follow-up Visit
Number analyzed (Participants) | 10 | 9
T-score
  Physical T-Score | 35.5 (5.70) | 33.96 (4.24)
  Mental T-Score | 43.02 (4.17) | 40.52 (7.26)

20. Secondary Outcome: Frequency of Rescue Medication Use
Description: The opioid sparing effect of NAS ketamine will be determined by evaluating frequency of rescue medications use prior to and during the study.
Time Frame: Visit 1 through Visit 5, up to 6 weeks
Population: Due to inconsistencies with participant-reported pill counts, the data for rescue medication use could not be reliably analyzed.
Arm/Group | Intranasal Ketamine Treatment
Number analyzed (Participants) | 0

21. Secondary Outcome: Total Opioid Consumption
Description: The opioid sparing effect of NAS ketamine will be determined by evaluating total opioid consumption (rescue medication) prior to and during the study.
Time Frame: Visit 1 through Visit 5, up to 6 weeks
Population: Due to inconsistencies with participant-reported pill counts, the data for total opioid consumption use could not be reliably analyzed.
Arm/Group | Intranasal Ketamine Treatment
Number analyzed (Participants) | 0

22. Post Hoc Outcome: Systolic Blood Pressure
Description: Blood pressure was measured at Baseline and up to 240 minutes after administration of ketamine.
Time Frame: Baseline, Minutes 5, 10, 15, 30, 45, 60, 120, 180, 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
millimeters of mercury (mmHg)
  Baseline | 118.6 (19.7) | 117.5 (20.8) | 117.6 (20.0) | 115.8 (19.3)
  Minute 5 | 117.8 (19.2) | 134.4 (30.7) | 119.9 (20.0) | 118.3 (14.8)
  Minute 10 | 122.3 (19.0) | 129.6 (23.3) | 122.9 (20.2) | 120.2 (19.1)
  Minute 15 | 119.0 (23.0) | 124.0 (20.9) | 123.1 (25.0) | 123.1 (16.9)
  Minute 30 | 121.7 (22.0) | 117.2 (20.6) | 125.4 (23.0) | 124.9 (18.1)
  Minute 45 | 119.8 (22.3) | 117.4 (15.1) | 121.3 (18.5) | 117.0 (18.4)
  Minute 60 | 116.9 (19.4) | 114.1 (13.4) | 118.7 (20.8) | 118.6 (17.4)
  Minute 120 | 117.2 (18.9) | 111.5 (13.4) | 114.9 (17.8) | 111.5 (13.0)
  Minute 180 | 111.9 (24.7) | 115.9 (15.5) | 116.3 (19.3) | 111.7 (13.2)
  Minute 240 | 116.2 (23.4) | 111.7 (12.9) | 118.2 (19.4) | 116.5 (23.9)

23. Post Hoc Outcome: Diastolic Blood Pressure
Description: Blood pressure was measured at Baseline and up to 240 minutes after administration of ketamine.
Time Frame: Baseline, Minutes 5, 10, 15, 30, 45, 60, 120, 180, 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
mmHg
  Baseline | 72.5 (7.2) | 76.3 (10.7) | 73.5 (9.8) | 72.2 (9.0)
  Minute 5 | 73.0 (9.1) | 82.4 (11.0) | 72.1 (9.4) | 74.4 (10.1)
  Minute 10 | 76.6 (7.9) | 81.1 (6.4) | 75.2 (9.8) | 73.2 (11.8)
  Minute 15 | 73.4 (6.8) | 78.5 (6.3) | 74.1 (10.6) | 76.8 (8.3)
  Minute 30 | 74.3 (6.7) | 72.2 (8.1) | 75.9 (11.2) | 77.1 (8.6)
  Minute 45 | 74.8 (7.4) | 71.7 (12.3) | 75.5 (10.8) | 73.4 (8.8)
  Minute 60 | 73.0 (7.3) | 73.6 (6.3) | 75.4 (11.3) | 73.4 (10.5)
  Minute 120 | 72.9 (8.9) | 72.9 (7.3) | 72.1 (7.5) | 72.2 (8.1)
  Minute 180 | 69.1 (11.1) | 71.9 (6.1) | 69.0 (6.5) | 70.8 (10.0)
  Minute 240 | 73.3 (7.32) | 70.2 (5.5) | 72.7 (6.4) | 75.3 (11.9)

24. Post Hoc Outcome: Heart Rate
Description: Heart rate was measured at Baseline and up to 240 minutes after administration of ketamine.
Time Frame: Baseline, Minutes 5, 10, 15, 30, 45, 60, 120, 180, 240, during Study Visits 1 through 4, up to 4 weeks
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine
Number analyzed (Participants) | 10 | 10 | 10 | 10
beats per minute
  Baseline | 80.0 (19.6) | 82.2 (18.4) | 81.3 (16.0) | 79.5 (14.6)
  Minute 5 | 80.4 (19.6) | 84.3 (18.2) | 76.7 (14.2) | 79.9 (13.6)
  Minute 10 | 78.9 (17.0) | 81.1 (15.2) | 75.7 (12.7) | 79.7 (14.5)
  Minute 15 | 77.3 (15.4) | 78.4 (16.2) | 76.6 (13.0) | 81.6 (15.5)
  Minute 30 | 79.1 (17.2) | 75.3 (13.2) | 74.2 (12.0) | 81.2 (16.4)
  Minute 45 | 78.7 (17.7) | 73.2 (17.5) | 75.2 (12.0) | 79.7 (15.0)
  Minute 60 | 75.9 (16.5) | 74.4 (14.2) | 75.8 (13.6) | 80.3 (16.0)
  Minute 120 | 81.6 (18.7) | 78.5 (17.9) | 76.1 (16.2) | 78.9 (15.9)
  Minute 180 | 79.1 (20.4) | 76.7 (15.6) | 78.0 (16.7) | 80.0 (16.0)
  Minute 240 | 80.9 (21.6) | 80.2 (17.8) | 74.0 (13.6) | 79.8 (14.2)

ADVERSE EVENTS:
Time Frame: Data collection for adverse events began at the first study visit and were followed by a telephone call 14 days after the last dose of study medication administration, up to 6 weeks.
Groups:
- Phone Call 14 Days Post-Last Dose: Participants were called 14 days after the last dose of study medication to assess adverse events.
Arm/Group | 10 mg Intranasal Ketamine | 10 mg Intravenous (IV) Ketamine | 30 mg Intranasal Ketamine | 50 mg Intranasal Ketamine | Follow-up Visit | Phone Call 14 Days Post-Last Dose
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10 | 2/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10 | 9/10 | 8/10 | 5/10 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg Intranasal Ketamine (N=10) | 10 mg Intravenous (IV) Ketamine (N=10) | 30 mg Intranasal Ketamine (N=10) | 50 mg Intranasal Ketamine (N=10) | Follow-up Visit (N=10) | Phone Call 14 Days Post-Last Dose (N=10)
Abdominal pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Neck tumor swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg Intranasal Ketamine (N=10) | 10 mg Intravenous (IV) Ketamine (N=10) | 30 mg Intranasal Ketamine (N=10) | 50 mg Intranasal Ketamine (N=10) | Follow-up Visit (N=10) | Phone Call 14 Days Post-Last Dose (N=10)
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0
Blurry vision (Eye disorders) | 1 | 2 | 1 | 1 | 0 | 0
Burning sensation in nostril (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Change in hearing (Ear and labyrinth disorders) | 0 | 2 | 0 | 1 | 0 | 0
Change in sense of smell (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Diaphoresis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 0
Dizziness (General disorders) | 1 | 6 | 3 | 4 | 0 | 0
Drowsiness (General disorders) | 2 | 1 | 1 | 3 | 0 | 0
Euphoria (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Facial numbnes (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Facial warmth (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 0 | 0 | 0
Feeling of unreality (General disorders) | 1 | 6 | 3 | 1 | 1 | 0
Floating sensation (General disorders) | 0 | 1 | 1 | 1 | 0 | 0
Foul taste (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Fuzzy thinking (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 2 | 2 | 4 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 1 | 0 | 0 | 0
In touch with emotions (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mood change (Psychiatric disorders) | 0 | 2 | 1 | 2 | 0 | 0
Nausea (General disorders) | 1 | 4 | 1 | 2 | 0 | 0
Night sweats (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0
Nightmares (General disorders) | 0 | 1 | 1 | 1 | 0 | 0
Restlessness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Somnolence (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Tongue numbness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision changes (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0
Visual hallucination (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intermittent nose bleeds (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT03146806/Prot_SAP_000.pdf